CLINICAL TRIAL: NCT02438566
Title: Non-inferiority Trial of Oral Tranexamic Acid (OTA) vs. Intravenous Tranexamic Acid (IVTA) to Prevent Blood Loss in Joint Replacement Surgery
Brief Title: Non-inferiority Trial of Oral Tranexamic Acid vs. Intravenous Tranexamic Acid in Joint Replacement Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The New England Baptist Hospital (Other)
Responsible Party: Principal Investigator, Kenneth Bauer, Principal Investigator, The New England Baptist Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 654455
Record Dates: First submitted 2015-04-14; First posted 2015-05-08 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis; Blood Loss, Surgical; Blood Loss, Postoperative
Keywords: Tranexamic Acid; Blood Loss; Total Hip Replacement; Bilateral Knee Replacement
MeSH Terms: conditions — Osteoarthritis; Blood Loss, Surgical; Postoperative Hemorrhage; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Tranexamic Acid (OTA) (Active Comparator): Subjects will be randomized 1:1 to receive either IVTA or OTA with corresponding placebos. OTA will be given as 1950 mg 1-2 hours prior to OR and 1950 mg 2 hours after surgical close, before discharge from PACU.
  Interventions: Drug: Tranexamic Acid (Oral)
- Intravenous Tranexamic Acid (IVTA) (Active Comparator): Subjects will be randomized 1:1 to receive either IVTA or OTA with corresponding placebos. IVTA will be given as 1 g intravenously at time of first incision (THA or bTKA without tourniquet) or just before 1st tourniquet application (bTKA), and then again, 1 g after final surgery closure.
  Interventions: Drug: Tranexamic Acid (Intravenous)

INTERVENTIONS:
Drug: Tranexamic Acid (Oral) — OTA will be given as 1950 mg 1-2 hours prior to OR and 1950 mg 2 hours after surgical close, before discharge from PACU.
  Other Names: trans-4-(aminomethyl)cyclohexanecarboxylic acid; Lysteda
  Arms: Oral Tranexamic Acid (OTA)
Drug: Tranexamic Acid (Intravenous) — IVTA will be given as 1 g intravenously at time of first incision (THA or bTKA without tourniquet) or just before 1st tourniquet application (bTKA), and then again, 1 g after final surgery closure.
  Other Names: trans-4-(aminomethyl)cyclohexanecarboxylic acid; Cyklokapron
  Arms: Intravenous Tranexamic Acid (IVTA)

SUMMARY:
The purpose of this research is to determine if the oral form of a medication (tranexamic acid) to reduce bleeding can be used in place of an intravenous (IV) form, to learn the best way to give tranexamic acid: either a pill by mouth, or a solution by vein.

DETAILED DESCRIPTION:
The purpose of this research is to determine if the oral form of a medication (tranexamic acid) to reduce bleeding can be used in place of an intravenous (IV) form.to learn the best way to give tranexamic acid: either a pill by mouth, or a solution by vein. Tranexamic acid is a medicine that reduces blood loss and reduces the need for blood transfusions in surgery. This drug is not experimental and has been used widely to treat patients in many settings, including orthopedic procedures, to reduce bleeding. This medication is now part of the standard of care at many centers in the U.S. and around the world. Orthopedic procedures have used iv tranexamic acid more often, but there are reasons to believe that the oral form may be at least equivalent and perhaps better at lower cost to the health care system. No other study has yet performed a systematic comparison to answer the question.

ELIGIBILITY:
Inclusion Criteria:

* To be included into this study, you must be undergoing hip or bilateral knee replacement surgery.
* You must be healthy enough to undergo joint replacement surgery.
* You must be able to understand and sign an informed consent.
* You must be at least 18 years of age.

Exclusion Criteria:

* You cannot be under 18 years of age.
* You cannot be undergoing revision hip or revision bilateral knee replacement surgery.
* You cannot be part of this study if you are allergic to the medication
* You cannot participate if you are on hemodialysis,
* You cannot participate if you have active coronary artery disease and if you have various vascular stents in place.
* You will also be excluded if you have ever had a blood clot (deep vein thrombosis (DVT), pulmonary embolism (PE)).
* You will also be excluded if you have ever had a cerebral or subarachnoid hemorrhage (brain bleeding), or stroke (cerebral vascular accident or transient ischemic attack).
* If you are on estrogen-containing medication (hormone replacement therapy or oral contraceptive) within 7 days of surgery, you cannot take part in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Lower number of units of blood required for transfusion. | 2 Years
  Lower number of units of blood required for transfusion in the OR and post-operatively, hospital-wide.

SECONDARY OUTCOMES:
Lower incidences of patients requiring blood transfusion. | 2 Years
  Lower incidences of patients requiring blood transfusion in the OR, or post-operatively.
Lower Blood Loss in Patients | Hospital Stay: 1-3 days.
  Lower amounts of blood loss in patients during in surgery, and post-operatively.
Length of Stay | 1-3 Days
  Potential for a shorter length of hospital stay for post-surgical patients.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Bauer, MD, Principal Investigator — New England Baptist Hospital
Locations (1):
- New England Baptist Hospital, Boston, Massachusetts, United States